CLINICAL TRIAL: NCT04197453
Title: The Cardiovascular Multi-dimensional Observational Investigation of the Use of PCSK9 Inhibitors (cvMOBIUS)
Acronym: cvMOBIUS
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Amgen (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20180059
Record Dates: First submitted 2019-12-05; First posted 2019-12-13 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: ASCVD
Keywords: Lipids; Lipid-lowering therapy; Coronary heart disease; Peripheral arterial disease; Proprotein convertase subtilisin/kexin type 9 inhibition; Effectiveness
MeSH Terms: conditions — Coronary Disease; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Consented Arm: Subjects with a recent (within 18 months) hospitalization for myocardial infarction, unstable angina, ischemic stroke, or critical limb ischemia, and subjects undergoing coronary, peripheral, or carotid revascularization, including surgical and percutaneous revascularization, with an LDL-C greater than or equal to 70 mg/dL who may be eligible for PCSK9 inhibitor therapy.
- Electronic Health Record (EHR) arm: Subjects with an inpatient or outpatient diagnosis of clinical ASCVD within the prior 12 months including coronary heart disease, ischemic cerebrovascular disease, atherosclerotic peripheral arterial disease, or prior coronary or peripheral or carotid revascularization.

SUMMARY:
cvMOBIUS is a North American registry of patients with ASCVD aimed at understanding patterns of care in ASCVD while evaluating the real world effectiveness of PCSK9 inhibitors.

DETAILED DESCRIPTION:
The purpose of this registry is to evaluate the effectiveness of proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors (PCSK9i) to reduce cardiovascular events among subjects presenting with a recent atherosclerotic cardiovascular disease (ASCVD) event in real-world practice. A total of 8500 patients with a recent cardiovascular event who are likely to be eligible for non-statin lipid lowering therapy will be enrolled and followed prospectively for five years. In addition, the study will assess longitudinal patterns of lipid control, clinical outcomes, and LLT including statins, ezetimibe, and PCSK9 inhibitors in adults with an ASCVD event and/or revascularization. This study will also compare the clinical characteristics and outcomes of subjects enrolled in both arms of the registry to understand the strengths and limitations of data harvested directly from electronic health record (EHR) systems as compared with prospectively collected information.

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥ 40 years
* One or both of the following:

  * Hospitalization for a clinical ASCVD event: acute (MI), UA, IS, or critical limb ischemia (CLI) within 18 months of enrollment NOTE: subjects must have been admitted to the hospital. Those who are admitted and discharged in less than 24 hours are eligible for the study. Subjects who have been admitted to the ER for a clinical ASCVD event and not admitted to the hospital are not eligible for enrollment.
  * Coronary, peripheral, or carotid revascularization including percutaneous or surgical revascularization in the past 18 months Note: Revascularization procedures can occur in the inpatient or outpatient setting.
* One of the following:

  * Low-density lipoprotein (LDL) ≥ 70 mg/dL (1.81 mmol/L) with no plans for immediate initiation or titration of statin therapy (Note: Subjects should not be enrolled into study during initiation/titration of statins until they have a stable LDL-C measurement > 4 weeks after their last statin change and no immediate plans for future titration).
  * Newly started on PCSK9i after the index hospitalization/procedure and prior to enrollment (but no more than 6 months prior to enrollment) with pre-PCSK9i treatment LDL-C value available and known background LLT any time prior to PCSK9i initiation.
* Planned follow-up within the health system.

Exclusion Criteria:

* Unable or unwilling to provide informed consent, including but not limited to cognitive or language barriers (reading or comprehension)
* Lack of phone or email for contact
* Evidence of end stage renal disease (ESRD) or stage 5 chronic kidney disease (CKD)
* Anticipated life expectancy less than 6 months
* On a PCSK9i prior to their qualifying event; Note: Subjects with prior PCSK9i use occurring and ending before the 12-month period prior to enrollment and before the index ASCVD event will be considered for inclusion.

EHR Arm Criteria:

Subjects are eligible to be included in the "EHR arm" of the registry if they are:

* Adults age ≥ 40 years of age
* Have at least 1 inpatient or outpatient diagnosis of clinical ASCVD within 12 months prior to enrollment including CHD, ischemic cerebrovascular disease, atherosclerotic PAD, or prior coronary or peripheral or carotid revascularization.

  * No exclusion criteria will be applied.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a recent ASCVD event or coronary, peripherial or carotid revascularization (in the prior 18 months).
  All subjects must have an LDL-C >=70 mg/dL or have initiated a PCSK9 inhibitor in the 6 months prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 752 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Incident event rate for the composite of all-cause mortality, non-fatal myocardial infarction (MI), and non-fatal ischemic stroke (IS). | Through study completion, a minimum of 4.5 years and maximum of 5 years
  Number of incident all-cause deaths, non-fatal MI, and non-fatal IS events (whichever occurs first) divided by the person-time at risk

SECONDARY OUTCOMES:
Incident event rate for all-cause mortality | Through study completion, a minimum of 4.5 years and maximum of 5 years
  Number of all-cause deaths divided by the person-time at risk
Incident event rate for non-fatal MI | Through study completion, a minimum of 4.5 years and maximum of 5 years
  Number of incident non-fatal MI events divided by the person-time at risk
Incident event rate for non-fatal IS | Through study completion, a minimum of 4.5 years and maximum of 5 years
  Number incident non-fatal IS events divided by the person-time at risk
Incident rate of coronary or peripheral or carotid revascularication procedures | Through study completion, a minimum of 4.5 years and maximum of 5 years
  Number of incident coronary or peripherial or carotid revascularization procedures
Incident event rate for major adverse limb events (MALE) including amputation | Through study completion, a minimum of 4.5 years and maximum of 5 years
  Number of incident MALE events divided by the person-time at risk. MALE is defined as the composite of ALI, major amputation (above the knee or below the knee, excluding forefoot or toe), or urgent revascularization (thrombolysis or urgent vascular intervention for ischemia).
Incident event rate for cardiovascular death | Through study completion, a minimum of 4.5 years and maximum of 5 years
  Number of cardiovascular deaths divided by the person-time at risk
Incident event rate for transient ischemic attack (TIA) | Through study completion, a minimum of 4.5 years and maximum of 5 years
  Number of incident TIA events divided by the person-time at risk
Incident event rate for unstable angina (UA) | Through study completion, a minimum of 4.5 years and maximum of 5 years
  Number of incident UA events divided by the person-time at risk
Longitudinal patterns of lipid control, use of and persistence with lipid lowering therapies (LLT) including statins, ezetimibe, and PCSK9 inhibitors | Through study completion, a minimum of 4.5 years and maximum of 5 years
  Describe patterns of lipid control and LLT's over time
The strengths and limitations of data harvested directly from electronic health record (EHR) systems as compared with prospectively collected information | Through study completion, a minimum of 4.5 years and maximum of 5 years
  Describe and compare clinical characteristics, ASCVD events, patterns of lipid control, and use of LLT's assessed via prospective data collection to those captured directly via an EHR data harvest.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (164):
- United States (143):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Old Pueblo Cardiology, Tucson, Arizona
  - Cardiovascular Research Foundation of Southern California, Beverly Hills, California
  - Los Alamitos Cardiovascular, Los Alamitos, California
  - Consortium of Attending Physicians for Research Investigations LLC, Los Angeles, California
  - Nanavati Critical Care Cardiology Clinic, National City, California
  - Rancho Cucamonga Clinical Trials, Rancho Cucamonga, California
  - Eisenhower Desert Cardiology Center, Rancho Mirage, California
  - San Diego Cardiac Center, San Diego, California
  - Millennium Clinical Trials, Thousand Oaks, California
  - Central Coast Cardiovascular, Ventura, California
  - University of Colorado Memorial Health System, Colorado Springs, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Cardiology Associates of Fairfield County, PC, Stamford, Connecticut
  - Bay Area Cardiology, Brandon, Florida
  - Holy Cross Hospital Inc, Fort Lauderdale, Florida
  - The Cardiac and Vascular Institute Research, Gainesville, Florida
  - Baptist Heart Specialists, Jacksonville Beach, Florida
  - Southwest Florida Research LLC, Naples, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Palm Harbor Medical Associates, Palm Harbor, Florida
  - Cardiology Consultants, Pensacola, Florida
  - Genesis Clinical Research Inc, Tampa, Florida
  - Interventional Cardiac Consultants, Trinity, Florida
  - Albany Internal Medicine, Albany, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Accel Research Sites, Atlanta, Georgia
  - First Georgia Physicians Group, Fayetteville, Georgia
  - Northwest Heart Clinical Research LLC, Arlington Heights, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Evanston Premier Healthcare Research LLC, Evanston, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Prairie Cardiovascular Consultants, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - Saint Vincent Heart Center, Indianapolis, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - MercyOne Iowa Heart Center, West Des Moines, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Premier Medical Group, Owensboro, Kentucky
  - Grace Research LLC, Bossier City, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Clinical Trials of America Inc, Monroe, Louisiana
  - University Medical Center-New Orleans, New Orleans, Louisiana
  - Ochsner Health Systems, New Orleans, Louisiana
  - Willis Knighton Cardiology, Shreveport, Louisiana
  - Grace Research LLC, Shreveport, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - MedStar Health Research Institute Chesapeake Cardiovascular Associates, Hyattsville, Maryland
  - TidalHealth Peninsula Regional, Inc, Salisbury, Maryland
  - McLaren Health, Bay City, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Jackson Heart, Jackson, Mississippi
  - Missouri Cardiovascular Specialists, Columbia, Missouri
  - University of Missouri Health Care, Columbia, Missouri
  - Cox Medical Centers, Springfield, Missouri
  - Washington University, St Louis, Missouri
  - Saint Louis Heart and Vascular PC, St Louis, Missouri
  - Methodist Physicians Clinic Heart Consultants, Omaha, Nebraska
  - Palm Research Center Inc, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Advanced Heart Care LLC, Bridgewater, New Jersey
  - Advanced Cardiology LLC, Cedar Knolls, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Virtua Health, Inc., Voorhees Township, New Jersey
  - Albany Medical College, Albany, New York
  - Bassett Healthcare, Cooperstown, New York
  - Long Island Cardiovascular Consultants, Lake Success, New York
  - SJH Cardiology Associates, Liverpool, New York
  - Winthrop University Hospital, Mineola, New York
  - Northwell Health, New York, New York
  - DiGiovanna Institute for Medical Education and Research, North Massapequa, New York
  - Circuit Clinic, Orchard Park, New York
  - Saratoga Clinical Research, LLC, Saratoga Springs, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefiore Medical Center - Bronx, The Bronx, New York
  - Duke Heart Center Clinical Research, Durham, North Carolina
  - Cone Health, Greensboro, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - Vidant Cardiology, Greenville, North Carolina
  - Novant Health Heart and Vascular Institute, Monroe, North Carolina
  - Coastal Carolina Health Care PA, New Bern, North Carolina
  - Pinehurst Medical Clinic, Inc, Pinehurst, North Carolina
  - WakeMed, Raleigh, North Carolina
  - Sanford Cardiology, Sanford, North Carolina
  - PMG Research of Piedmont HealthCare, Statesville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Premier Cardiovascular, Dayton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Heart House Research Foundation, Springfield, Ohio
  - Saint Vincent Medical Center, Toledo, Ohio
  - Central Oklahoma Early Detection Center, Edmond, Oklahoma
  - Ascension St John Clinical Research Institute, Tulsa, Oklahoma
  - Oklahoma State University Health Science Center, Tulsa, Oklahoma
  - Lynn Institute of Tulsa, Tulsa, Oklahoma
  - Central PA Physicians Group, Altoona, Pennsylvania
  - Capital Area Research LLC, Camp Hill, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Doylestown Health Cardiology, Doylestown, Pennsylvania
  - The Heart Group of Lancaster General Health, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Kent Hospital, Warwick, Rhode Island
  - AnMed Health, Anderson, South Carolina
  - PMG Research of Charleston, Charleston, South Carolina
  - Columbia Heart, Columbia, South Carolina
  - Upstate Cardiology, Greenville, South Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Diagnostic Cardiology Group, Chattanooga, Tennessee
  - Stern Cardiovascular Foundation Inc, Germantown, Tennessee
  - Parkway Cardiology Associates, Oak Ridge, Tennessee
  - Seton Heart Institute, Austin, Texas
  - Thyroid Endocrinology and Diabetes, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Northwest Houston Cardiology, Houston, Texas
  - North Dallas Research Associates, McKinney, Texas
  - CardioVoyage, McKinney, Texas
  - Texas Institute of Cardiology, McKinney, Texas
  - Southern Endocrinology Associates PA, Mesquite, Texas
  - Permian Research Foundation, Odessa, Texas
  - Consano Clinical Research, San Antonio, Texas
  - San Antonio Endovascular and Heart Institute, San Antonio, Texas
  - Village Medical Centers, The Woodlands, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Cardiology Consultants of Danville, Inc, Danville, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
  - Cardiovascular Associates of Virginia, Midlothian, Virginia
  - Tidewater Physicians Multispecialty Group Clinical Research, Newport News, Virginia
  - York Clinical Research LLC, Norfolk, Virginia
  - Multicare Institute for Research and Innovation, Puyallup, Washington
  - Washington University, Seattle, Washington
  - Marshall Cardiology, Huntington, West Virginia
  - West Virginia University, Morgantown, West Virginia
- Canada (21):
  - Fraser River Endocrinology, Surrey, British Columbia
  - Cardio Metabolic Collaborative Clinic, Victoria, British Columbia
  - Discovery Clinical Services Ltd, Victoria, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - South Sherbrook Health Centre and Pharmacy, Winnipeg, Manitoba
  - Cardio 1, Winnipeg, Manitoba
  - Brampton Clinical Trials, Brampton, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Saul Vizel Professional Medicine Corporation â€" Vizel Cardiac Research, Cambridge, Ontario
  - Cardiovasular Clinical Research Organization Limited, Greater Sudbury, Ontario
  - Curnew Medicine Professional Corporation, Hamilton, Ontario
  - Partners in Advanced Cardiac Evaluation, Newmarket, Ontario
  - Oakville Cardiovascular Research Limited Partnership, Oakville, Ontario
  - Rhema Research Institute, Owen Sound, Ontario
  - Heart Health Institute Research Incorporated, Scarborough Village, Ontario
  - Sewa Ram Singal Medicine Professional Corporation, Toronto, Ontario
  - Mohan Babapulle Medicine Professional Corporation, Waterloo, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - McGill University Health Centre - Montreal General Hospital, Montreal, Quebec
  - Applied Medical Informatics Research Incorporated, Montreal, Quebec
  - CardioVasc HR Incorporated, Saint-Jean-sur-Richelieu, Quebec

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com